CLINICAL TRIAL: NCT00946686
Title: A Relative Bioavailability, Parallel Study Of Leflunomide 20 mg Tablets Under Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability, Parallel Study Of Leflunomide 20 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B023709
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic | interventions — Leflunomide

ARMS (2):
- 1 (Experimental): Leflunomide 20 mg Tablets (Geneva Pharmaceutical)
  Interventions: Drug: Leflunomide 20 mg Tablets (Geneva Pharmaceutical)
- 2 (Active Comparator): Arava 20 mg Tablets (Aventis Pharmaceutical, Inc.)
  Interventions: Drug: Arava 20 mg Tablets (Aventis Pharmaceutical, Inc.)

INTERVENTIONS:
Drug: Leflunomide 20 mg Tablets (Geneva Pharmaceutical)
  Arms: 1
Drug: Arava 20 mg Tablets (Aventis Pharmaceutical, Inc.)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability, parallel study Of Leflunomide 20 mg tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-09; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services